CLINICAL TRIAL: NCT03168893
Title: Deep Brain Stimulation on the Subgenual Cingulate and Accumbens Nucleus for Patients With Chronic, Severe and Resistant Anorexia Nervosa
Brief Title: Deep Brain Stimulation for Patients With Chronic, Severe and Resistant Anorexia Nervosa
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Parc de Salut Mar (Other)
Responsible Party: Principal Investigator, Víctor Pérez, PhD MD, Parc de Salut Mar
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Treatment
Other Study IDs: ECP-AN-2016-01
Record Dates: First submitted 2017-05-25; First posted 2017-05-30 (Actual); Last update posted 2020-02-21 (Actual); Status verified 2020-02

CONDITIONS: Anorexia Nervosa
Keywords: deep brain stimulation
MeSH Terms: conditions — Anorexia Nervosa | interventions — Deep Brain Stimulation

STUDY DESIGN:
Who Masked: Participant, Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Deep brain stimulation ON (Experimental): Surgical procedure is necessary.In surgery, two cerebral electrodes (either in the Subgenual cingulate or in the Accumbens Nucleus) are connected to a subcutaneous generator at abdominal fat level, under general anesthesia. The patient will initiate the stimulation prior to discharge . At 6 months follow up, Deep brain stimulation continue 3 months more activated, patient and psychiatrist don´t know
  Interventions: Device: Deep brain stimulation ON
- Deep brain stimulation OFF (Experimental): Surgical procedure is necessary.In surgery, two cerebral electrodes (either in the Subgenual cingulate or in the Accumbens Nucleus) are connected to a subcutaneous generator at abdominal fat level, under general anesthesia. The patient will initiate the stimulation prior to discharge . At 6 months follow up, Deep brain stimulation is stopped during 3 months , patient and psychiatrist don´t know
  Interventions: Device: Deep brain stimulation OFF

INTERVENTIONS:
Device: Deep brain stimulation ON — Infinity model of deep brain stimulation is placed ( 2 brain elecrodes and subcutaneus generator ) under general anhestesia. The system is activated
  Other Names: Deep Brain Stimulation: Infinity model device (ON)
  Arms: Deep brain stimulation ON
Device: Deep brain stimulation OFF — Infinity model of deep brain stimulation is placed ( 2 brain elecrodes and subcutaneus generator ) under general anhestesia. The system is not activated
  Other Names: Deep Brain Stimulation: Infinity model device (OFF)
  Arms: Deep brain stimulation OFF

SUMMARY:
Deep brain stimulacion (DBS) clinical study in the subcallosal cingulate (CSG) and accumbens nucleus (NAc) for 8 patients with treatment-refractory, cronic and severe anorexia nervosa (AN) patients. The main objective is to show efficacy and safety. Studies show that SSG and NAc are strategical targets in the pathophysiology and the hypothetical surgical treatment in AN patients. The patients distribution (4 patients in each target) it will made by the AN type and the comorbidity associated, the reasons are: 1- It is well known the comorbidity treatment imoportance in the AN evolution, 2- The two differentes types of AN have differents clinical behaviour and prognosis, 3- Studies show efficacy in TOC and DM patients with NAc DBS and in DM patients with CSG DBS. The main variable is BMI. After a 6 months stabilization evaluation phase will be followed (only in patients that have increase 10% BMI) by a double-bind, crossover phase, where patients will receive 3 months with stimulation turned on and 3 month with turned off. All patients will have a 12 months follow up. The study secondary objectives are to know the relation btween the stimulacion answer (increase 10% BMI) and the differents variables, specially AN type, associated cormobidity, selected target and preoperative MRI tractography study.

DETAILED DESCRIPTION:
HYPOTHESIS OF THE CLINICAL TRIAL

Based on the results of functional, preclinical, clinical and neurocircuit imaging studies in patients with Anorexia Nervosa (AN) and in the results of deep brain stimulation (DBS) in 81 other mental illnesses and in AN, our main hypotheses are:

1. The subgeneric cingulate (CSG) and nucleus accumbens (NAc) are strategic targets in AN patients, so deep brain stimulation in these two targets may be effective in the treatment of AN patients.
2. The stimulation of the CSG and the NAc has been safe in other mental illnesses so it can also be in patients with AN.

VARIABLES

The variables to be studied are: age, years of illness, number of admissions, type of AN, drugs tested, drugs at the present time, non-pharmacological treatments received, weight and current BMI, weight and mean BMI of the last year, associated comorbidity, Hamilton Scale for Depression (HAMD-17), Hamilton Scale for Anxiety (HAMA), Obsessive Compulsive Yale-Brown Scale (YBOCS), Cornell Scale for Eating Disorder (YBC-EDS), Quality of Life Scale SF-36, stimulation variables (voltage, frequency, pulse amplitude, active contacts), stimulated target (CSG, NAc), complications.

The main variable is the Body Mass Index (BMI). The baseline will be the mean BMI of the last 3 months pre-dating.

The variables will be collected preoperatively, after the surgery on a monthly basis until the end of the 12 months of follow-up from the surgery, and in the last month of follow-up of the study (month 33 of the study). Patient visits will be every 2 weeks from the start of the stimulation to 12 months of follow-up.

Response and referral criteria. Response to treatment is considered if BMI increases at least 10% of baseline BMI (baseline BMI: the mean of the last 3 months pre-engagement). Remission is considered if the BMI is greater than 18.5. The type of response in the associated comorbidities will be studied as a variable, but not as a criterion of response to treatment.

Concomitant treatments during the study: Patients will continue with the pharmacological treatment and with the previous psychotherapeutic therapies. During the study, modification of the drugs will not be allowed, but a dose adjustment if not an increase of more than 50%. All this must be recorded on the data collection sheet in the usual way. A new psychotherapeutic therapy can not be initiated during the study, and if it is done, the patient would leave the study.

Rescue measures against side effects of stimulation. The complication rate is very low (1-4%). In case of an infectious complication, the patient will receive antibiotic treatment. In case of a neurological complication (comitial crisis, feeling of discomfort), the generator can be turned off and restarted once the complication is resolved.

Rescue measures if clinical worsening in the off phase of double-blind. The generator will be connected, and the patient leaves the double-blind phase.

Rescue measures if worsening AN or some of their comorbidities (patient under stimulation). Pharmacological dose adjustment is permitted if it is not an increase of more than 50%, in case of having to be done, the patient would leave the study. It would not be possible to initiate a psychotherapy in which the patient was no longer present and, if required, the patient would leave the study.

Criteria for modifying the stimulation variables. There are two criteria that can modify the stimulation parameters: that there is no response to treatment (BMI), or that there is a side effect related to the stimulation (for example, a crisis in the hospital, discomfort). Changes in patient comorbidity will not be a criterion for modifying pacing parameters.

STAGES OF THE STUDY

Stage 1 (Documentation and recruitment). Its duration is 3-6 months. At this stage, all necessary documentation will be processed and the patients included in the study will be recruited, following the inclusion and exclusion criteria described below.

Stage 2 (Preoperative Evaluation, Surgical Intervention and Follow-up). This stage comprises month 4 to month 33 of the study. Once the patient was included in the study, with confirmation of the evaluation committee, and having received informed consent of the patient, the preoperative evaluation will be performed (Brain Resonance with tensor tractography, general analysis, chest x-ray, Electrocardiogram, psychometric tests, weight, body mass index, and neuropsychological evaluation). The period for the surgical procedure comprises month 4 to month 22 of the study, since all patients will be evaluated during a follow-up period of at least 12 months, and after a follow-up period, a period of evaluation of the results (3 months) is required. All surgeries and follow-up will be performed at the Hospital del Mar. In surgery, two cerebral electrodes (either in the Subgenual cingulate or in the Accumbens Nucleus) are connected to a subcutaneous generator at abdominal fat level, under general anesthesia, the hospitalization time is 3-4 days. The patient will initiate the stimulation of the stimulation system implanted prior to discharge. The patient will have control visits every 2 weeks (face-to-face or telephone) and monthly at the Hospital del Mar for the evaluation of scales, weight and possible side effects during the study's duration (minimum 1 year per patient). The patient will undergo an intraoperative cerebral CT scan and an immediate postoperative CT scan. Neuropsychological evaluation will be performed preoperatively and after 6 months of treatment. The follow-up stage of the patients in the study comprised month 4 of the study and month 33 of the study.

Stage 3 (Double Blind). This stage comprises a period of 6 months. After 6 months of stimulation, patients responding to stimulation (10% or greater increase in BMI compared to the mean BMI of the last 3 months of pre-engagement) will go on to a double-blind phase, in which 3 Months in on and 3 months in off, or vice versa (assigned by envelopes prior to the start of surgeries). Those patients who are in the off and worsen group (5% decrease in BMI from baseline) will be rescued by reestablishing the stimulation, and leaving the cross-study phase.In order to preserve masking, the CoiP (neurosurgeon, responsible for programming), will decide the changes in the stimulation remaining unrelated to the evaluation of the patients.

Stage 4 (Total collection of data and conclusions). This stage comprises from month 34 to month 36 of the study (last month of the project's 3 years).

ELIGIBILITY:
Inclusion Criteria:

(All criteria for inclusion must be met)

1. Age between 18-60 years
2. Diagnosis of AN, both restrictive type and compulsion / purge type defined by the DSM-V-TR
3. Chronicity: minimum of 10 years of illness.
4. Resistance to treatment, shown by one or both of the following situations:

   A. That of the multiple treatments performed, at least 1 is an intensive treatment (hospitalization or day hospital), with one or more of the following results:
   * I have not been able to finish the treatment.
   * That it has finished but with little or no answer.
   * That in spite of having finished it, and of having answered, Has found a subsequent relapse in the first six months. B. Clinical situation of medical instability, accompanied by refusal to participate in any treatment program and including at least 1 episode of admission for involuntary feeding.
5. Extremely serious (BMI less than 15), or severe (BMI between 15-15,99)
6. Ability to sign informed consent
7. Ability to undergo all tests and follow-ups of the study

Exclusion Criteria:

1. BMI less than 13 at the time of recruitment for the study.
2. Psychosis in the present moment or in the past.
3. Current neurological disease.
4. Substance or alcohol abuse and dependence in the last year.
5. Contraindications to perform a brain MRI
6. Presence of cardiac arrhythmias or other cardiac, respiratory, renal or endocrine affections, as a result of AN or not, that carries risk for the surgical procedure.
7. Pregnancy

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 8 (Estimated)
Dates: Start 2017-05-23 (Actual); Primary Completion 2020-03-17 (Estimated); Study Completion 2020-12-17 (Estimated)

PRIMARY OUTCOMES:
Body mass index (BMI) | From baseline till 12 months
  BMI will be measured monthly from baseline till 12 months. Data will be compared with BMI in the beginning of the open label period

SECONDARY OUTCOMES:
Adverse events during the study | From baseline till 12 months
Psychiatric comorbidity | From baseline till 12 months
  Psychiatric comorbidity will be measured monthly from baseline till 12 months

CONTACTS AND LOCATIONS:
Overall Officials: Gloria Villalba Martínez, Doctor, Study Director — Parc de Salut Mar
Locations (1):
- Gloria Villalba Martinez, Barcelona, Spain

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Hayes DJ, Lipsman N, Chen DQ, Woodside DB, Davis KD, Lozano AM, Hodaie M. Subcallosal Cingulate Connectivity in Anorexia Nervosa Patients Differs From Healthy Controls: A Multi-tensor Tractography Study. Brain Stimul. 2015 Jul-Aug;8(4):758-68. doi: 10.1016/j.brs.2015.03.005. Epub 2015 May 21. PMID 26073966
- [Result] Cleary DR, Ozpinar A, Raslan AM, Ko AL. Deep brain stimulation for psychiatric disorders: where we are now. Neurosurg Focus. 2015 Jun;38(6):E2. doi: 10.3171/2015.3.FOCUS1546. PMID 26030702
- [Result] Lipsman N, Lozano AM. Targeting emotion circuits with deep brain stimulation in refractory anorexia nervosa. Neuropsychopharmacology. 2014 Jan;39(1):250-1. doi: 10.1038/npp.2013.244. No abstract available. PMID 24317325
- [Result] Lipsman N, Woodside DB, Giacobbe P, Lozano AM. Neurosurgical treatment of anorexia nervosa: review of the literature from leucotomy to deep brain stimulation. Eur Eat Disord Rev. 2013 Nov;21(6):428-35. doi: 10.1002/erv.2246. Epub 2013 Jul 19. PMID 23873668
- [Result] Sun B, Liu W. Stereotactic surgery for eating disorders. Surg Neurol Int. 2013 Apr 17;4(Suppl 3):S164-9. doi: 10.4103/2152-7806.110668. Print 2013. PMID 23682343
- [Result] Oudijn MS, Storosum JG, Nelis E, Denys D. Is deep brain stimulation a treatment option for anorexia nervosa? BMC Psychiatry. 2013 Oct 31;13:277. doi: 10.1186/1471-244X-13-277. PMID 24175936
- [Result] Treasure J, Ashkan K. Deep brain stimulation for anorexia nervosa: a step forward. Eur Eat Disord Rev. 2013 Nov;21(6):507-8. doi: 10.1002/erv.2253. Epub 2013 Sep 20. No abstract available. PMID 24115472
- [Result] Lipsman N, Woodside B, Lozano AM. Evaluating the potential of deep brain stimulation for treatment-resistant anorexia nervosa. Handb Clin Neurol. 2013;116:271-6. doi: 10.1016/B978-0-444-53497-2.00022-X. PMID 24112901
- [Result] Benabid AL. Comment on 'Treatment of intractable anorexia nervosa with inactivation of the nucleus accumbens using stereotactic surgery'. Stereotact Funct Neurosurg. 2013;91(6):373. doi: 10.1159/000348279. Epub 2013 Oct 9. No abstract available. PMID 24108085
- [Result] Lipsman N, Woodside DB, Lozano AM. Deep brain stimulation for anorexia nervosa - authors' reply. Lancet. 2013 Jul 27;382(9889):306. doi: 10.1016/S0140-6736(13)61631-1. No abstract available. PMID 23890039
- [Result] McLaughlin NC, Didie ER, Machado AG, Haber SN, Eskandar EN, Greenberg BD. Improvements in anorexia symptoms after deep brain stimulation for intractable obsessive-compulsive disorder. Biol Psychiatry. 2013 May 1;73(9):e29-31. doi: 10.1016/j.biopsych.2012.09.015. Epub 2012 Nov 3. No abstract available. PMID 23128051
- [Result] Wu H, Van Dyck-Lippens PJ, Santegoeds R, van Kuyck K, Gabriels L, Lin G, Pan G, Li Y, Li D, Zhan S, Sun B, Nuttin B. Deep-brain stimulation for anorexia nervosa. World Neurosurg. 2013 Sep-Oct;80(3-4):S29.e1-10. doi: 10.1016/j.wneu.2012.06.039. Epub 2012 Jun 25. PMID 22743198
- [Derived] Perez V, Villalba-Martinez G, Elices M, Manero RM, Salgado P, Gines JM, Guardiola R, Cedron C, Polo M, Delgado-Martinez I, Conesa G, Medrano S, Portella MJ. Cognitive and quality-of-life related factors of body mass index (BMI) improvement after deep brain stimulation in the subcallosal cingulate and nucleus accumbens in treatment-refractory chronic anorexia nervosa. Eur Eat Disord Rev. 2022 Jul;30(4):353-363. doi: 10.1002/erv.2895. Epub 2022 Mar 23. PMID 35322504